CLINICAL TRIAL: NCT05913180
Title: Vitamin C for the Prevention of Catheter-associated Urinary Tract Infections in Women Who Undergo Elective Gynecological Surgeries: a Randomized Double-blinded Controlled Trial
Brief Title: Vitamin C Effectiveness in Preventing Urinary Tract Infections After Gynecological Surgeries
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Collaborators: Moscow State University of Medicine and Dentistry (Other)
Responsible Party: Principal Investigator, Tony Bazi, Associate Professor of Clinical Obstetrics and Gynecology, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 62/137-H/77-2023-25-2295
Record Dates: First submitted 2023-06-10; First posted 2023-06-22 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Catheter-Associated Urinary Tract Infection
Keywords: Ascorbic acid; Vitamin C; Elective Gynecologic surgeries; CAUTI
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin C (Active Comparator): 1000mg Ascorbic acid daily starting the day of elective gynecological surgery for 10 days
  Interventions: Drug: Ascorbic Acid 1000 MG
- Placebo (Placebo Comparator): Placebo daily starting the day of elective gynecological surgery for 10 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ascorbic Acid 1000 MG — 1000mg Ascorbic acid orally daily started on the day of elective gynecological surgery for 10 days
  Other Names: Vitamin C
  Arms: Vitamin C
Drug: Placebo — Placebo tablet daily starting day of elective gynecological surgery for 10 days
  Arms: Placebo

SUMMARY:
Double-blind placebo-controlled randomized trial aiming to assess the role of Vitamin C supplementation in the prevention of catheter-associated urinary tract infections in women undergoing elective gynecological surgeries.

DETAILED DESCRIPTION:
Women undergoing Elective GYN surgery are a particularly high-risk group for UTIs, because these operations involve surgery adjacent to the bladder and delayed bladder emptying is common. It has been estimated that the 'risk of Urinary tract infections among women undergoing elective Gynecologic GYN surgery is between 10-64%, following catheter removal. Catheterization, in itself, poses a significant risk for UTIs because insertion and removal introduce bacteria and cause trauma, both of which may increase the risk of UTIs. The incidence of UTI for women in the general population is estimated to be 3-4% per year vs 5% per day of catheterization. For this reason, multiple interventions have been studied for the prevention of UTIs. Ascorbic acid (vitamin C) is often suggested as a supplement that can prevent recurrent UTIs by acidification of the urine. Strong clinical evidence to support this claim in healthy adult women is lacking. Because of the lack of literature regarding the use of Vitamin C as a prophylactic agent for the prevention of UTIs, the investigators wish to conduct this study to assess the potential therapeutic efficacy of Ascorbic acid in preventing UTIs after elective GYN surgery.

ELIGIBILITY:
Inclusion Criteria:

* Nonpregnant women
* 18 years of age or older
* Undergoing elective GYN surgery

Exclusion Criteria:

* Pregnant women
* Already taking Vitamin C supplementation
* Nephrolithiasis
* Congenital anomaly or neurogenic bladder
* Allergy to ascorbic acid
* On therapeutic anticoagulant medicine during the 6 weeks after surgery
* Gynecological surgery involving fistula repair or a vaginal mesh removal
* Positive Urinalysis in the pre-admission unit
* Recurrent UTIs
* Diabetes
* G6PD
* Hemochromatosis
* Renal disorders

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 180 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of UTI | 30 days
  The Primary endpoint is the proportion of participants who experience a clinically diagnosed and treated UTI as evidenced by a positive urine culture.

SECONDARY OUTCOMES:
Asymptomatic UTI | 30 days
  The proportion of participants with a positive urine culture, while asymptomatic (asymptomatic bacteriuria) at the end of the study period

CONTACTS AND LOCATIONS:
Overall Officials: Tony Bazi, M.D., Principal Investigator — American University of Beirut Medical Center
Locations (1):
- Moscow State University of Medicine and Dentistry, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foxman B, Cronenwett AE, Spino C, Berger MB, Morgan DM. Cranberry juice capsules and urinary tract infection after surgery: results of a randomized trial. Am J Obstet Gynecol. 2015 Aug;213(2):194.e1-8. doi: 10.1016/j.ajog.2015.04.003. Epub 2015 Apr 13. PMID 25882919
- [Background] Ochoa-Brust GJ, Fernandez AR, Villanueva-Ruiz GJ, Velasco R, Trujillo-Hernandez B, Vasquez C. Daily intake of 100 mg ascorbic acid as urinary tract infection prophylactic agent during pregnancy. Acta Obstet Gynecol Scand. 2007;86(7):783-7. doi: 10.1080/00016340701273189. PMID 17611821
- [Background] Carlsson S, Wiklund NP, Engstrand L, Weitzberg E, Lundberg JO. Effects of pH, nitrite, and ascorbic acid on nonenzymatic nitric oxide generation and bacterial growth in urine. Nitric Oxide. 2001 Dec;5(6):580-6. doi: 10.1006/niox.2001.0371. PMID 11730365
- [Background] Trautner BW, Darouiche RO. Catheter-associated infections: pathogenesis affects prevention. Arch Intern Med. 2004 Apr 26;164(8):842-50. doi: 10.1001/archinte.164.8.842. PMID 15111369
- [Background] Barbosa-Cesnik C, Brown MB, Buxton M, Zhang L, DeBusscher J, Foxman B. Cranberry juice fails to prevent recurrent urinary tract infection: results from a randomized placebo-controlled trial. Clin Infect Dis. 2011 Jan 1;52(1):23-30. doi: 10.1093/cid/ciq073. PMID 21148516
- [Background] Hickling DR, Nitti VW. Management of recurrent urinary tract infections in healthy adult women. Rev Urol. 2013;15(2):41-8. PMID 24082842
- [Background] Wald HL, Ma A, Bratzler DW, Kramer AM. Indwelling urinary catheter use in the postoperative period: analysis of the national surgical infection prevention project data. Arch Surg. 2008 Jun;143(6):551-7. doi: 10.1001/archsurg.143.6.551. PMID 18559747